CLINICAL TRIAL: NCT02688244
Title: Randomized Trial Comparing Irrigation Versus Suction in Laparoscopic Appendectomy for Complicated Acute Appendicitis in Adults
Brief Title: Irrigation Versus Suction in Complicated Acute Appendicitis
Acronym: ISAAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Jesus Abrisqueta Carrion, PhD, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAC-2015-HCUVA
Record Dates: First submitted 2015-12-01; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Appendicitis; Abdominal Abscess; Acute Disease; Cecal Diseases; Infection
Keywords: complicated appendicitis; laparoscopic appendectomy; irrigation; suction; abdominal abscess
MeSH Terms: conditions — Appendicitis; Abdominal Abscess; Acute Disease; Cecal Diseases; Infections | interventions — Therapeutic Irrigation; WASH protein, Drosophila; Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irrigation (Active Comparator): Irrigation of the area with at least 300ml normal saline using the power suction/irrigator
  Interventions: Procedure: Irrigation
- No irrigation (Active Comparator): Only suction with the power suction/irrigator without saline attached
  Interventions: Procedure: No irrigation

INTERVENTIONS:
Procedure: Irrigation — Irrigation of the abdominal cavity with at least 300ml of normal saline using the power suction/irrigator
  Other Names: Washout
  Arms: Irrigation
Procedure: No irrigation — Suction only, using suction device
  Other Names: Suction
  Arms: No irrigation

SUMMARY:
This study evaluates the intraabdominal abscess rate after laparoscopic appendectomy in complicated acute appendicitis performing irrigation of the abdominal cavity or only suction without lavage.

DETAILED DESCRIPTION:
Despite the available literature for and against the irrigation of the abdominal cavity in complicated acute appendicitis, in the current practice of this and other centres, the irrigation and no irrigation is made equally depending on the surgeon who performs the intervention.

Those who systematically irrigate the abdominal cavity in laparoscopic appendectomies do it as an inherited act from open surgery and those who systematically do not irrigate the abdominal cavity base their choice in theories such as abscess migration due to the irrigation and difficulty of the suction of all the irrigated fluid, spreading, therefore, the infection.

The intention of the investigators is to provide evidence about this technique in order to either systematize peritoneal irrigation in laparoscopic appendectomy for complicated appendicitis or avoid an unnecessary gesture, if it were established so.

This will be a prospective, randomized clinical trial involving patients who present to the hospital with complicated acute appendicitis. Power calculation was based on abscess rate in the investigators' hospital calculated retrospectively (15%) Subjects will be those patients above 18 y.o. who are found to have complicated acute appendicitis (defined as perforated appendicitis before or during surgery, gangrenous appendicitis and/or purulent peritonitis).

The final decision to include a patient in the study will made after complication has been visually confirmed during surgery. The randomization assignment will be made known at the initiation of the operation, and confirmation of complication will confirm the patient will utilize the next randomization slot.

The irrigation group will have suction irrigator set up with a 1 liter bag of normal saline. The surgeon must use at least 300 ml of this bag but may use as much as they choose.

The no irrigation group will have the suction irrigator set up without the saline attachment. This will leave them with the capacity for suction only. Since several suction devices exist, this will assure the same type of suction for both groups.

After the operation, both groups will be managed in the same manner. When the patient is tolerating a regular diet, on oral pain medication and has been afebrile for over 12 hours, they will be discharged on oral antibiotics to complete a course of 7 days. If the participants stay until the 5th post-operative day, a white blood cell count will be checked, which if it is normal, they will be discharged to home without antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complicated acute appendiccitis
* Laparoscopic approach

Exclusion Criteria:

* Open approach
* Medical or psychiatric condition of the patient that compromises the informed consent authorisation
* Non complicated acute appendicitis
* Underage patients (<18)
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative abscess | 1 month
  Number of post-operative abscesses in each arm
Location of post-operative abscess | One month
  Number of abscesses in every quadrant of the abdomen
Treatment of post-operative abscess | One month
  Number of post-operative abscesses treated with a radiological drain

SECONDARY OUTCOMES:
Operating time | 1 day
  Length of surgery, in minutes.
Hospital stay (Time until discharge) | 2 weeks
  Time until discharge, in days.
Postoperative pain (Visual analogic scale) | 6 days
  Visual analogic scale, from 1 to 10
Postoperatory fever | 6 days
  Body temperature in Celsius degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de La Arrixaca, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided